CLINICAL TRIAL: NCT02820558
Title: A Phase I Study of Safety and Pharmacological Activity of Substance P (sP) in the Reversal of Recent-Onset Type 1 Diabetes (T1D)
Brief Title: Neuropeptide Therapy of Recent Onset Type 1 Diabetes
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vanilloid Genetics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VanilloidGenetics-001-13
Record Dates: First submitted 2016-05-19; First posted 2016-07-01 (Estimated); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Neuropeptide; Therapy; Onset
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Substance P

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Substance P - 1nmol/kg (Experimental): Substance P 1nmol/kg intra-celiac artery, single treatment
  Interventions: Drug: Substance P
- Substance P - 5nmol/kg (Experimental): Substance P 5nmol/kg intra-celiac artery, single treatment
  Interventions: Drug: Substance P
- Substance P - 15nmol/kg (Experimental): Substance P 15nmol/kg intra-celiac artery, single treatment
  Interventions: Drug: Substance P
- Substance P - 45nmol/kg (Experimental): Substance P 45nmol/kg intra-celiac artery, single treatment
  Interventions: Drug: Substance P

INTERVENTIONS:
Drug: Substance P

SUMMARY:
This study evaluates the delivery of substance P via the celiac artery in the treatment of recent onset type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Recent onset T1D (CDA 2013 guidelines: See link in links section
* Age 10-18 years
* Disease Duration 3-30 months
* Fasting C-Peptide (measured at screening) greater than or equal to 33 pmol/L
* Post honeymoon phase based on the following criteria: History of HbA1c values and insulin requirements from diagnosis indicating a honeymoon period followed by increased insulin requirements which at time of recruitment are > 0.50 units/Kg together with an HbA1c value > 7.2 %; Patients with diabetes duration > 3 months who never experienced a honeymoon period as reflected by consistent HbA1c values > 7.2 % from the time of diagnosis and at the time of recruitment are using an insulin dose > 0.50 units/Kg.
* The presence of one or more of the TRPV1 alleles similar to those found in patients currently enrolled in the TRPV1-North American - European Study.
* Stimulated C-Peptide (measured at mixed meal tolerance at Stage A and Stage B of sP trial) ≥ 200 pmol/L and less than or equal to 1500 pmol/L.

Exclusion Criteria:

* Patients with known co-morbidities, including ACE-inhibitor treated hypertension as well as chromosomal abnormalities, involving one or more organ systems.
* Type 2 Diabetes Mellitus
* Patients with a known radiographic contrast allergy
* Pregnancy.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 2016-05; Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Stage A Safety: Side effects reported for entire cohort | Reported during the first 20-27 days following sP administration
  To determine if there are unexpected adverse events with intra arterial delivery of sP into the celiac artery in individuals with Type 1 Diabetes, and evidence of residual beta cell function as reflected by a peak C---peptide levels of > 200 pmol/L. Multiple measurements per patient will be aggregated to arrive at one reported value: Number of participants with abnormal laboratory values, adverse events and/or peak C-peptide levels >200pmol/L that are related to treatment.

SECONDARY OUTCOMES:
C-Peptide Levels (small cohort) | Day 20-27 post sP injection
  To determine in an initial small cohort (n=12, toxicity and dose finding cohort) if one or more sP doses significantly increases the basal or stimulated c---Peptide levels at Day 20---27 post---injection using data from Mixed Meal Tolerance Test (MMTT).
C-Peptide Levels (large cohort) | Day 20-27 post sP injection
  To assess in a larger cohort (n=40, continued safety and efficacy) whether sP dose, determined from the dose finding cohort, significantly increases basal or stimulated C-- peptide levels at Day 20---27 post sP---injection using MMTT data.

OTHER OUTCOMES:
sP Longevity | 3 and 6 months
  To determine an estimate of sP longevity in the entire cohort of patients, by monitoring HbA1c values, exogenous insulin requirement, daily recorded blood sugar levels and adverse event recording at 3 and 6 months post injection of sP. Multiple measurements per patient will be aggregated to arrive at one reported value for the aforementioned outcome measures.

CONTACTS AND LOCATIONS:
Overall Officials: Etienne Sochett, MD, Principal Investigator — Hospital for Sick Children, Toronto Ontario
Locations (1):
- Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- See also: CDA 2013 guidelines — http://guidelines.diabetes.ca/Browse/Chapter3